CLINICAL TRIAL: NCT05954832
Title: Changes in Loading Conditions on Induction of General Anesthesia: Mechanisms of Post-Induction Hypotension (PIH)
Brief Title: A Study of Changes in Heart Function and Blood Flow in People Receiving Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-079
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia
Keywords: Changes in Heart Function; Changes in Blood Flow; Echocardiography; 23-079
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Echocardiography: Patients participating in this study will undergo routine anesthetic and perioperative care with the addition of an echocardiography and Clearsight BP measurement.
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography and Clearsight BP measurements before, immediately after anesthesia induction and after intubation (for 20 min)

SUMMARY:
The purpose of this study is to understand changes in heart function (how the heart pumps blood) and blood flow in people who receive general anesthesia during surgery. The researchers are particularly interested in the heart function and blood flow changes in people who experience low blood pressure (hypotension) after receiving anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age requiring general anesthesia for surgery
* Intubation required for anesthetic management / surgery
* Anticipated prep time before incision of 20 minutes
* Baseline MAP >70mmHg

Exclusion Criteria:

* History of coronary artery disease
* History of cardiac disease (e.g., HTN, arrythmias, valvular and structural abnormalities)
* History of peripheral artery occlusive disease
* Beta-blocker use
* Anti-hypertensive medication use
* Patients with epidural, spinal, paravertebral, serratus blocks preoperatively
* Patients requiring rapid sequence induction (where intubation occurs concurrently with induction)
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring general anesthesia for surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with post-induction hypotension (PIH) | up to 20-mins after anesthesia induction.
  summarize the distributions of the echocardiography parameter values (pre-load LVEDd(cm), after-load LVEDs(cm), other measures [e.g., contractility (EF %) and structural abnormalities]) across each timepoint among patients with and without PIH

CONTACTS AND LOCATIONS:
Overall Officials: Anahita Dabo-Trubelja, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm